CLINICAL TRIAL: NCT03735329
Title: Polso SpO2 Accuracy Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChroniSense Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR 2018-307
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2018-11

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pulse oximetry monitoring (Experimental)
  Interventions: Device: Diagnostic test of SPO2

INTERVENTIONS:
Device: Diagnostic test of SPO2 — The SpO2 accuracy of the test devices will be evaluated over the oxygen saturation range between 70-100%.

SUMMARY:
The purpose of this study is to validate the oxygen saturation (SpO2) accuracy of the Polso Monitoring System during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry for SpO2 validation

DETAILED DESCRIPTION:
The purpose of this study is to validate the SpO2 accuracy and performance of the Polso Monitoring System during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry for SpO2 validation. It is expected that the Accuracy Root Mean Square (Arms) performance of the Polso Monitoring System will meet a specification of 3.5% or less in non-motion conditions for the range of 70-100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

The Control Pulse Oximeter, an FDA cleared device, is used to monitor the oxygen saturation levels real time throughout the study for subject safety and to target stable plateaus. This device is used to assess the stability of the data.

A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.

A minimum of 10 healthy adult subjects, ranging in pigmentation from light to dark, will be enrolled in the study to meet the study design requirements defined by ISO 80601-2-61:2011 and by the FDA's Guidance for Pulse Oximeters. The subjects will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels.

The study population will include 10-15 healthy non-smoking (or has refrained from smoking for 2 days) competent adults 18-50 years of age. The subject selection will be an equitable distribution of males and females of any race with varying skin tones including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger. Data collection will occur over a 2-5 day period for this study population.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 4 males and a minimum of 4 females, with the balance made up of either
* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* Smoker Subjects who have refrained will be screened for COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery with continued indications of health issues ,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen).
  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months)
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with severe allergies to iodine (only applicable if iodine or similar is used)
* Subjects with severe allergies lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio < 0.4)
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
SpO2 percentage | Through study completion, 1 month average
  Percentage of SpO2 measured by the Polso Monitoring System during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. Data analysis will follow ISO80601-2-61, Annex EE and the FDA Guidance Document for Pulse Oximeters (March 4, 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Avista Adventist Hospital, Staff Anesthesiologist
Locations (1):
- Clinimark Desaturation Laboratory, Site ID# 001, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No